CLINICAL TRIAL: NCT05009342
Title: Evaluation of Functional Outcomes at 2 Months According to Therapeutic Management, in Trauma With Low-grade Osteo-ligamentous Ankle Injury in Children
Acronym: CHEVIPED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of patients very limited due to lack of time and human resources dedicated to research.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29BRC21.0016
Record Dates: First submitted 2021-08-06; First posted 2021-08-17 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-07

CONDITIONS: Ankle Injuries; Ligament Injury
Keywords: low-grade; osteo-ligament injuries; children; soft resin ankle brace; Below-knee rigid resin cast
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, non-inferiority, without blinding, controlled trial with 2 parallel groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Below-knee soft resin cast (Experimental): Below-knee soft resin cast is administered to participants in emergency department. Investigator puts three layers of jersey supplemented by strips of soft resins to be unrolled along the leg after immersion in warm water
  Duration to ankle immobilization with soft resin boot : 21 days.
  Interventions: Device: below-knee soft resin cast
- Below-knee rigid resin cast (Other): Below-knee soft resin cast is administered to participants in emergency department. Investigator puts one layer of jersey and then one layer of foam composed by strips of cotton wool to be unrolled supplemented by strips of rigid resins to be unrolled along the leg after immersion in warm water.
  Duration to ankle immobilization with soft resin boot : 21 days.
  Interventions: Device: Below-knee rigid resin cast

INTERVENTIONS:
Device: below-knee soft resin cast — Patients have soft resin boot between day 0 (inclusion visit) and day 21 (follow-up visit n°1)
  Arms: Below-knee soft resin cast
Device: Below-knee rigid resin cast — Patients have rigid resin boot between day 0 (inclusion visit) and day 21 (follow-up visit n°1)
  Arms: Below-knee rigid resin cast

SUMMARY:
Lack of current consensus on the therapeutic management of low-grade osteo-ligament injuries in ankle trauma in children. Several types of immobilization are evaluated in the literature, with different conclusions. Some teams recommend a functional treatment similar to the adult (with or without strict immobilization), others remain on standard rigid immobilizations.

The goal of the study is to simplify and homogenize the therapeutic management of low-grade osteo-ligament injuries in ankle trauma in children.

DETAILED DESCRIPTION:
Lack of current consensus on the therapeutic management of low-grade osteo-ligament injuries in ankle trauma in children. Several types of immobilization are evaluated in the literature, with different conclusions. Some teams recommend a functional treatment similar to the adult (with or without strict immobilization), others remain on standard rigid immobilizations.

The goal of the study is to simplify and homogenize the therapeutic management of low-grade osteo-ligament injuries in ankle trauma in children.

CHEVIPED is a controlled, randomized, comparative monocentric trial.

Randomization into 2 groups and stratified on presence to fracture Salter 1 and age

Experimental group : Patients with below-knee soft resin cast Control group : Patients with below-knee rigid resin cast.

The primary objective is to demonstrate at 2 months that with post traumatic low- grade osteo-ligamentous ankle injury the recovery of physical function are at least as effective with a below-knee soft resin cast compared to a below-knee rigid resin cast.

The secondary objectives are :

1. Clinical evaluation of treatment at 3 weeks in immediate post-immobilization.
2. Evaluation of the management satisfaction (effectiveness and understanding) and the treatment tolerance .
3. Evaluation of the time taken to resume painless support after immobilization.
4. Point of interest evaluation
5. Determine the diagnostic performance of the "combined clinical criteria" in comparison with the ultrasound/radiography couple.
6. Evaluation of the diagnostic performance of clinical inspection criteria (edema, bruise) in high-grade ligament damage.
7. Evaluation of the link between the "combined clinical criteria" and the results of the radiography.
8. Evaluation of the relationship between "combined clinical criteria" and ultrasound results.
9. Evaluation of the link between the results of radiography and ultrasound.

200 patients are expected to be included.

Inclusion period : 12 months. Duration of patient's participation: 2 months Total study duration: 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Walking child from 5 to 15 years old.
* From hour 0 to hour 48 of ankle trauma with torsion mechanism (inversion, eversion or rotation).
* Patient presenting for the first time to the emergency room for this traumatic episode.
* Possibility of carrying out an ultrasound during the passage to the emergency room.
* Child and parents' consent in the study participation

Exclusion Criteria:

* Pubescent patients requiring anticoagulation (menarche in girls and genital pilosity in boys).
* Direct shock on the foot without sprain mechanism.
* Fracture with deformation or open fracture.
* History of ankle trauma in the last 3 months.
* Neurological or neuromuscular pathology.
* Child with a delay in acquisitions and / or psychomotor development (difficulties in understanding and interacting to locate pain).
* Absence of a representative of parental authority.
* Constitutional bone disease or connective tissue.
* Acquired or congenital coagulopathy.
* Patient presenting beyond 48h of trauma.
* Polytraumatized.
* Dermabrasion, wound or sign of skin suffering next to the ankle requiring specific monitoring.
* Child or parents refusal in study participation

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Activities Scale for Kids (ASKp) | At 2 months
  Activities Scale for Kids (ASKp) is a questionnaire about activities from the previous week. It has 30 item with 5 answers : all of the time (the better) / most of the time / sometimes / once in a while / none of the time (the worse).

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | day 0
  It is a scale that measures pain intensity with small ruler, between 0 (no pain) to 10 (severe pain). It can be administered for children 4 to 6 years old.
Visual Analogue Scale (VAS) | day 21
  It is a scale that measures pain intensity with small ruler, between 0 (no pain) to 10 (severe pain). It can be administered for children 4 to 6 years old.
Numeric Scale (NS) | day 0
  It is a scale that mesures pain intensity. Children aged to 4 to 6 years gives a grade between 0 (no pain) to 10 (severe pain)
Numeric Scale (NS) | day 21
  It is a scale that measures pain intensity. Children aged to 4 to 6 years gives a grade between 0 (no pain) to 10 (severe pain)
Clinical exams | day 0
  Clinical exams are exams administered by investigator during a consultation. There are four exams :
  1. inspection : presence or not of a hematoma and oedema
  2. palpation : pain or not with palpation
  3. mobilization : 3 items with 2 answers (Yes/No)
  4. support capacity : 2 items with 2 answers (Yes/No)
Clinical exams | day 21
  Clinical exams are exams administered by investigator during a consultation. There are four exams :
  1. inspection : presence or not of a hematoma and oedema
  2. palpation : pain or not with palpation
  3. mobilization : 3 items with 2 answers (Yes/No)
  4. support capacity : 2 items with 2 answers (Yes/No)
Parents questionnaire | day 21
  It is a questionnaire for parents that assesses the feeling about the children care, with 3 questions.
Intercurrent consultation | between day 0 and day 42
  Adjudicated intercurrent consultation (Other medical consultation than those planned) during the study treatment period
injury during removal of the device | between day 0 and day 42
  Adjudicated injury during removal of the device during the study treatment period
Negative predictive value (VPN) of "combined clinical criteria" | day 0
  Negative predictive value (VPN) of "combined clinical criteria" in the detection of low-grade bone or ligament damage to the ankle in children compared to ultrasound/radiography.
Sensitivity and specificity of local skin signs | day 0
  Sensitivity and specificity of local skin signs (INSPECTION line of the clinical examination questionnaire) to detect high-grade ligament damage on ultrasound.
Comparison between clinical exams and the radiography results. | day 0
  Clinical exams are exams administred by investigator during a consultation (inspection, palpation, mobilization, support capacity).The results of this exams are compared to radiography results at the inclusion (origin and localization of injury)
Comparison between the clinical exams and the ultrasound results. | day 0
  Clinical exams are exams administred by investigator during a consultation (inspection, palpation, mobilization, support capacity).The results of this exams are compared to ultrasound results at the inclusion (origin and localization of injury) .
Comparison between the radiography results and the ultrasound results. | day 0
  Ultrasound results are compared to radiography results at the inclusion (origin and localization of injury) .

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.